CLINICAL TRIAL: NCT04214756
Title: Methodist Acute Pancreatitis Protocol
Acronym: MAPP
Status: Active, not recruiting | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 035.GID.2014.D
Record Dates: First submitted 2019-08-12; First posted 2020-01-02 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-04

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients treated pre-MAPP: The registry will collect data on all AP patients since August 2011, and will continue until a sufficient number of cases are obtained to reach statistical significance
- Patients treated post-MAPP: The registry will collect data on all AP patients since August 2011, and will continue until a sufficient number of cases are obtained to reach statistical significance
  Interventions: Procedure: Acute Pancreatitis

INTERVENTIONS:
Procedure: Acute Pancreatitis — All patients diagnosed with acute pancreatitis beginning August 2011 at MDMC, MCMC, MMMC, and MRMC will be included in the registry for analysis of baseline and clinical outcomes data and subsequently divided into two groups (i.e. those treated pre-MAPP and post-MAPP).
  Groups: Patients treated post-MAPP

SUMMARY:
The overall goal of this ongoing registry study is to optimize initial evaluation and treatment of patients with AP according to recommended guidelines, the Methodist Acute Pancreatitis Protocol (MAPP), which were implemented in January 2015.

DETAILED DESCRIPTION:
1.1. Background

Acute pancreatitis (AP) represents a significant burden for patients, their caregivers, and our healthcare delivery systems. The most common discharge gastrointestinal diagnosis is AP and more than two billion dollars is spent annually for management thereof . Costs are certainly even higher as the incidence of AP has increased. Admit frequency for AP doubled in 15 years before 2002 such that more than 200,000 admissions were attributed to AP, and the trend toward increased admissions for AP has continued. Overall, about 20% of AP cases are severe and the risk for fatality attributed to severe AP is significant (> 25%). Classification of AP severity is defined into three groups: mild, moderately severe, and severe. These categories have been validated in that standard clinical outcomes correlate well with the severity of AP.

There are several principle gaps in knowledge with respect to AP. First, it remains challenging to initially predict the ultimate severity of acute pancreatitis . Some patients presenting with what is thought to be a mild attack of AP ultimately progress to having more severe disease. This is of utmost importance because outcomes of AP seem to be clearly related to very early diagnosis and appropriate initial management. For example, both morbidity and mortality for AP are closely related to persistent organ failure, which in theory might be prevented with very early appropriate management. It is also not clear if the existing data regarding prognostic scoring systems were influenced by early interventions. Secondly, we lack confirmatory data that following recommended guidelines for management of AP in fact results in improved clinical outcomes. It has been suggested that the care of AP patients has changed considerably during the last decade. One might assume that this change was in response to following one or all of several different guidelines produced by international societies. However, there is a paucity of outcomes data, particularly related to patients that have been cared for according to the recommended guidelines, and further investigation is warranted. Lastly, many AP studies include patients who had onset of symptoms more than several days prior to admission or transfer to a tertiary center; careful study is warranted in AP patients who present within one to two days of symptom onset.

The evaluation and treatment of all patients with AP according to specific guidelines embodies the principles of patient-centeredness research and improved clinical outcomes may also translate into better quality of life. Patients who suffer from severe AP that is complicated by pancreatic necrosis continue to have poor physical components of quality of life. However, the burden for patients with AP extends beyond the obvious clinical outcomes. Even as symptom scales from quality of life instruments improve following recovery, mental component scores remain significantly impaired.

1.2. AIMS/OBJECTIVES

Specific aims:

Aim 1: Compare the outcome of AP between the two groups. The total length of hospital stay (including ward stay and ICU stay) and the Discharge status (discharged or died) will be considered as the outcome of AP.

Aim 2: Compare the imaging study and hospital resource utilization (charges) between the two groups

Aim 3: Determine if the existing prognostic scoring systems are valid in this patient population when managed according the recommended guidelines.

1.3. HYPOTHESIS 1.4.1. Primary Hypothesis: The total length of hospital stay will be shorter for the group of patients treated after January 2015 (post-MAPP) than those treated before December 2014 (pre-MAPP). Additionally, more patients treated according to the guidelines will be discharged home (and not die in the hospital) as compared to the patients not treated according to the guidelines.

1.4.2. Secondary Hypothesis: There will be less utilization of imaging studies for patients treated according to the guidelines.

2.1. STUDY OBJECTIVES 2.1.1. Primary Objective Compare the total length of hospital stay (including ward stay and ICU stay) and the discharge status (discharged or died) between the pre- and post-MAPP AP patients.

2.1.2. Secondary Objectives

* Compare the imaging study and hospital resource utilization (charges) between the pre- and post-MAPP AP patients.
* Determine if the existing prognostic scoring systems are valid in the AP patient population when managed according the recommended guidelines

  3. STUDY DESIGN The proposed ongoing registry study will follow the cohort study design where baseline patient data and clinical outcomes data will be collected retrospectively. The registry will collect data on all AP patients since August 2011, and will continue until a sufficient number of cases are obtained to reach statistical significance. Retrospective data will be collected on patients diagnosed with AP based on two groups (those treated pre-MAPP and post-MAPP). Initial clinical criteria will be evaluated for the predictive value of AP severity in both groups.

  4. STUDY SETTING/LOCATION The study will be conducted with data from Methodist Dallas Medical Center (MDMC), Methodist Charlton Medical Center (MCMC), Methodist Mansfield Medical Center (MMMC) and Methodist Richardson Medical Center (MRMC).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Presented to ER with Acute severe pain for < 48 hours before presentation.
* Laboratory values of Lipase and/or amylase > 3X normal

Exclusion Criteria:

* History of recent penetrating or blunt abdominal trauma
* Patients transferred to MDMC for upper abdominal pain consistent with pancreatic etiology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with acute pancreatitis beginning August 2011 at MDMC, MCMC, MMMC, and MRMC will be included in the registry for analysis of baseline and clinical outcomes data and subsequently divided into two groups (i.e. those treated pre-MAPP and post-MAPP).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-04-05 (Actual); Primary Completion 2025-04-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Length of Hospital Stay | From April 2016 until Jun 2025 (anticipated study close)
  Length of hospital stay will be calculated in days with a discrete variable as [(discharge date - Admission date)].
Ward days | From April 2016 until Jun 2025 (anticipated study close)
  Length of ward days will be calculated in days with a discrete variable as [(discharge date from ward - Admission date to the ward)].
ICU days | From April 2016 until Jun 2025 (anticipated study close)
  Length of ICU stay will be calculated in days with a discrete variable as [(discharge date from ICU - Admission date to the ICU)].
Discharge status | From April 2016 until Jun 2025 (anticipated study close)
  will be recorded as a categorical variable indicating whether the discharge was to the home, SNF or rehab facility (1=Home; 2 = SNF; 3 = Rehab)

SECONDARY OUTCOMES:
CT scan | From April 2016 until Jun 2025 (anticipated study close)
  will be recorded as a binary variable indicating whether the CT scan was done in the ER (1 = Yes; 0 = No).
Empiric antibiotics | From April 2016 until Jun 2025 (anticipated study close)
  will be recorded as a binary variable indicating whether antibiotics were used (1 = Yes; 0 = No).
Harmless AP score (HAPS) | From April 2016 until Jun 2025 (anticipated study close)
  The Harmless Acute Pancreatitis Score is used to predicts within 30 minutes of admission patients whose acute pancreatitis will run a mild course. Scored from 0-4. A score of 0 is associated with the absence of pancreatic necrosis , and 4 with severe presence (Balthazar score, 0-4 points)
bedside index for severity in AP (BISAP) | From April 2016 until Jun 2025 (anticipated study close)
  Predicts mortality risk in pancreatitis, and is scored from 0 to 5. Patients with a BISAP Score of 0 would have <1% risk of mortality, whereas a score of 5 would indicate a mortality rate of 22%.
C reactive protein | From April 2016 until Jun 2025 (anticipated study close)
  C reactive protein levels produced in patient's liver would be evaluated
Procalcitonin | From April 2016 until Jun 2025 (anticipated study close)
  Procalcitonin levels produced in patients will be evaluated
organ dysfunction scores | From April 2016 until Jun 2025 (anticipated study close)
  organ dysfunction scores is scored from 0 to 5. If no organ dysfunction is present, the score is 0, rising to a maximum of 5.
Severity of acute pancreatitis (AP) | From April 2016 until Jun 2025 (anticipated study close)
  Severity of AP will be measured by categorizing into mild, moderately severe and severe according to the revised Atlanta classification (RAC).(7, 27) Mild severity is defined as having no organ failure and no local (acute fluid collection, acute necrotic collection, pseudocyst, walled-off necrosis) or systemic (exacerbation of preexisting co- morbidities) complications. Moderately severe AP is defined as transient organ failure (<48 hours) and/or local/systemic complications without persistent organ failure. And severe AP is defined as persistent single or multiple organ failure (> 48 h) (1= Mild; 2= Moderate severity; 3 = Severe AP). (27)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Tarnasky, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Methodist Health System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No